CLINICAL TRIAL: NCT05259176
Title: Effects of Transcranial Direct Current Electrical Stimulation (tDCS) on the Recovery of Ideomotor Apraxia of the Upper Limbs in Patients With Acute Stroke
Brief Title: Effects of Transcranial Direct Current Electrical Stimulation on the Recovery of Ideomotor Apraxia of the Upper Limbs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica di Riabilitazione Toscana Spa (Other)
Collaborators: FONDAZIONE GIANFRANCO SALVINI ONLUS (Unknown)
Responsible Party: Principal Investigator, CRISTIANO SCARSELLI, Deputy Chief Health Officer, Clinica di Riabilitazione Toscana Spa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: tDCS-AIM
Record Dates: First submitted 2022-02-15; First posted 2022-02-28 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Apraxia, Ideomotor
Keywords: transcranial direct current stimulation; stroke rehabilitation
MeSH Terms: conditions — Apraxia, Ideomotor | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The present study will be conducted in 2 recruiting centers with a randomized double-blind design. Post-stroke patients with apraxia will be randomly allocated into two parallel groups (Group A and Group B) by creating two randomisation lists of 10 patients which will allow for random and balanced assignment of patient numbers to either Group A or Group B. Group A will undergo direct current transcranial stimulation (tDCS) for 10 consecutive days and online treatment with Smania training. Group B will undergo sham stimulation for 10 consecutive days and online treatment with Smania training.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcranial Direct Current Stimulation (tDCS) (Experimental): transcranial Direct Current Stimulation (tDCS) on the left posterior parietal cortex and rehabilitative treatment with Smania's training
  Interventions: Device: transcranial Direct Current Stimulation (tDCS); Device: Behavioural
- Placebo stimulation (sham-tDCS) (Sham Comparator): Placebo stimulation and rehabilitative treatment with Smania's training
  Interventions: Device: Sham stimulation (sham-tDCS); Device: Behavioural

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — Direct current transcranial stimulation will be applied for 20 minutes over the left posterior parietal cortex with an intensity set to 2 mA.
  Arms: transcranial Direct Current Stimulation (tDCS)
Device: Sham stimulation (sham-tDCS) — The same positioning of electrodes as the stimulation condition will be used, but the current will be applied for 30 seconds and then progressively reduced.
  Arms: Placebo stimulation (sham-tDCS)
Device: Behavioural — Treatment for upper limbs ideomotor apraxia (Smania et al., 2000)

SUMMARY:
Limbs apraxia is a motor disorder whose characteristic is the inability or difficulty to perform intentional movements of the limbs (gestures), most frequently involving the upper limbs. Recent literature indicated promising effects of transcranial direct current stimulation (tDCS) in the recovery of limbs apraxia, showing that, in stroke patients, excitatory anodal tDCS over left inferior parietal lobe (IPL) may improve limb apraxia. Despite this encouraging evidence, the need for larger well powered and sham-controlled clinical trials has also been identified. For these reasons, the objective of this study is to investigate the effects of tDCS application on the left posterior parietal cortex, associated with the treatment for apraxia made by Smania et al. in 2000, on the recovery of the upper limbs ideomotor apraxia in patients with left brain lesion of vascular origin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both gender, with ischaemic stroke;
* Left hemispheric injury documented by neuroimaging examination;
* Cerebrovascular disease onset within the first 30 days;
* Presence of ideomotor apraxia as documented by a score < 53 in the De Renzi's test;
* Intact semantic skills as documented by normal performance on the Auditory or Visual Word Comprehension subtest of the Neuropsychological Examination for Aphasia (E. N. P. A.);
* Full comprehension skills as documented by normal performance in the sub-test of oral or orthographic comprehension (Auditory or Visual Words Comprehension) of the Neuropsychological Examination for Aphasia (E. N. P. A.);
* Age between 20 and 80 years;
* Any schooling;
* Patient's informed consent signature.

Exclusion Criteria:

* Comprehension and/or semantics deficit as documented by E. N. P. A.;
* Pre-existing psychiatric and/or neurological pathology;
* Failure to sign the patient's and/or caregiver's informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline Ideomotor apraxia test | The first day of treatment; End of 2nd week; End of 3rd week
  It consists of 24 imitation tests carried out with the fingers, the hand and the limb homolateral to the lesion.
  Each gesture is presented up to three times if the production is incorrect, and receives a score of 3 to 0 depending on whether the copy is correct the first, the second, the third time, or never. The test includes 24 gestures, 12 symbolic and 12 non-symbolic, for a total score of 72. Application of the test to over 200 normal subjects showed that the diagnosis of apraxia can be made reliably when the score drops below 53, it's probable, but not certain, for a score between 53 and 62, and it's excluded when the score is greater than 62.
Changes from baseline Standardized test for the diagnosis of a selective ideomotor apraxia deficit on the basis of gesture and effector types | The first day of treatment; End of 2nd week; End of 3rd week
  Test for ideomotor apraxia assessment which allows to highlight: 1) the selective deficits for the type of gesture to be imitated and, therefore, specific damage to the two processes underlying the imitation (direct route and semantic pathways) presenting known and new gestures in separate blocks; and 2) deficits of the distal or proximal component of the movements.
Changes from baseline Ideational apraxia test | The first day of treatment; End of 2nd week; End of 3rd week
  By placing in front of the patient one object at a time, he is asked to perform the pantomime of use of the object without touching or holding the object itself, but only by looking at it (visual mode). The examiner will assign 2 points if the execution is correct, 1 point if the execution is correct after repetition of the command and 0 points for always incorrect execution. The objects used are: glass, screwdriver, comb, gun, fork, key, rubber, saw, hammer, fan.

SECONDARY OUTCOMES:
Changes from baseline Oral apraxia test | The first day of treatment; End of 2nd week; End of 3rd week
  The examiner mimics the 10 bucco-facial movements required by the protocol, and asks the patient to imitate them. If the subject does not perform the task or does not perform it correctly, the therapist repeats the gesture a second time. If, again, the patient does not perform or makes a mistake, the next stimulus is taken. Maximum time for each stimulus is 30 seconds. The gestures to imitate are: show your tongue, whistle, yawn, try to lick your nose, make a partridge, give a kiss, show how your teeth shake when it's cold, snap your tongue making the sound of a galloping horse, blow and scratch your throat. The score is 2 if the execution is accurate on the first attempt, 1 if it is correct on the second attempt and 0 if the gesture is not executed or is not reproduced correctly.
Changes from baseline Jebsen-Taylor Hand Functional Assessment Scale | The first day of treatment; End of 2nd week; End of 3rd week
  It is a scale that allows to assess the level of hand function during daily activities. It consists of 7 subtests: writing, turning a page, lifting small objects, pantomime of eating, stacking objects, lifting large and light objects and large and heavy objects. The non-dominant hand will be tested first and then the dominant one. The time for each item will be timed: the final score (total time) will be given by the sum of all the part times: the lower the score, the better the level of hand function.

CONTACTS AND LOCATIONS:
Overall Officials: CRISTIANO SCARSELLI, Principal Investigator — Clinica di Riabilitazione Toscana Spa
Locations (1):
- CLINICA DI RIABILITAZIONE TOSCANA Spa, Montevarchi, Arezzo, Italy

IPD SHARING:
Plan to Share IPD: No